CLINICAL TRIAL: NCT04390828
Title: Effectiveness of Guided Imagery Meditation in Patients With Laparoscopic Gallstone Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ju Lu, Principal Investigator, National Yang Ming Chiao Tung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYMUH-IRB No. 2019A020
Record Dates: First submitted 2019-12-05; First posted 2020-05-18 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Gallstone
Keywords: Guided imagery meditation, Gallstones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery Meditation (Experimental): the guided image meditation invention program of the intervention measures of this study include four important elements: 1) Meditation exercises: the exercises to adjust the body and mind through specific attention, so that people gradually feel the state of relaxation through practice; (2) Guided image: the simple visualization and use of mental images produced by imagination as a form of psychotherapy, images come from natural scenes (e.g., forests and mountains, streams and oceans), positive feelings and emotions are generated through psychological imagination to induce psychological and physiological relaxation state; (3) Music aids: reaching a relaxed state with comfortable and slow background music; (4) Breathing relaxation training: the patient is taught to take abdominal breathing to divert attention and stimulate the parasympathetic nervous system to achieve muscle relaxation. The entire intervention process takes about 15 to 20 minutes, 2 times a day.
  Interventions: Behavioral: Guided Imagery Meditation
- Usual care (No Intervention): usual care

INTERVENTIONS:
Behavioral: Guided Imagery Meditation — the guided image meditation invention program of the intervention measures of this study include four important elements: 1) Meditation exercises: the exercises to adjust the body and mind through specific attention, so that people gradually feel the state of relaxation through practice; (2) Guided image: the simple visualization and use of mental images produced by imagination as a form of psychotherapy, images come from natural scenes (e.g., forests and mountains, streams and oceans), positive feelings and emotions are generated through psychological imagination to induce psychological and physiological relaxation state; (3) Music aids: reaching a relaxed state with comfortable and slow background music; (4) Breathing relaxation training: the patient is taught to take abdominal breathing to divert attention and stimulate the parasympathetic nervous system to achieve muscle relaxation. The entire intervention process takes about 15 to 20 minutes, 2 times a day.
  Arms: Guided Imagery Meditation

SUMMARY:
Guided image meditation has been shown to alter the functional circuits of the brain to alleviate pain by mediating breathing and thoughts. Therefore, the purpose of this study is to investigate whether the intervention with guided image meditation after laparoscopic cholecystectomy can effectively alleviate postoperative pain, reduce anxiety, promote sleep quality, and increase pain control satisfaction for the patients with gallstones.

DETAILED DESCRIPTION:
Gallstone is the most common digestive tract disease in general surgical wards. The incidence of gallstones in Chinese is about 5-10%, and the patients often seek hospital treatment due to abdominal pain. At present, most gallstones are treated with laparoscopic cholecystectomy, and postoperative pain is one of the most troublesome problems for surgical patients. However, up to 90% of patients undergoing abdominal surgery still experience moderate to severe pain, which not only affects the patient's physical recovery, but also causes psychological anxiety. Therefore, it is important to provide good postoperative pain management. Guided image meditation has been shown to alter the functional circuits of the brain to alleviate pain by mediating breathing and thoughts. Therefore, the purpose of this study is to investigate whether the intervention with guided image meditation after laparoscopic cholecystectomy can effectively alleviate postoperative pain, reduce anxiety, promote sleep quality, and increase pain control satisfaction for the patients with gallstones.

This study used 2×2 pre-test and post-test randomized control tests with randomized, single-blind, experimental study design. The research subjects were recruited from the general surgical ward of the North District Teaching Hospital. The study questionnaire included the assessment of pain levels using the 11-point Numeric Rating Scale (NRS-11) and the 11-face Face Pain Scale (FPS-11), the degree of anxiety using the Chinese version of Beck Anxiety Inventory (BAI), pain control satisfaction using Visual Analogue Scales (VAS), and sleep quality using the Chinese Pittsburgh Sleep Quality Index (CPSQI). The number of samples in this study was calculated by G-Power 3.1.2 statistical software. At least 68 samples were collected and grouped by random allocation, with 34 each for the control group (conventional scheme) and the experimental group (guided image meditation intervention). After the pre-test, the two groups were post-tested on the first postoperative day. The data obtained in this study were statistically analyzed by statistical software SPSS 22.0 for descriptive statistics including number of assignments, percentage, mean, standard deviation, Maximum and Minimum. Inferential statistical analysis by analysis of variance (ANOVA), Chi-square test, independent sample t-test, logistic regression, Pearson's correlation, repeated measures ANOVA and Generalized Estimating Equation (GEE) tested the pre-test and post-test results of the experimental group and the control group to compare the difference between the two groups in pain index, anxiety level, sleep quality and pain control satisfaction.

This study intended to use the characteristics of the guided image meditation being easy to learn and easy to operate and the evidence-based measures to alleviate postoperative pain, reduce anxiety, promote sleep quality and improve post-surgical pain control satisfaction to prove the empirical effect of guided image meditation in clinical care. It is hoped to provide an empirically based interventional effect to improve the problems associated with patients after laparoscopic surgery and improve the quality of life of patients after surgery. The results of this paper are expected to be published in domestic and foreign journals, so as to add to empirical academic literature and to be shared by medical staff for increasing new knowledge.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years old, and diagnosed as having gallstones and had laparoscopic cholecystectomy
* conscious, can communicate in Mandarin and Taiwanese; and have agreed to participate in the study.

Exclusion Criteria:

* with hearing or vision severely impaired
* cognitive mental disorder, such as mental illness
* who are unwilling to participate in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
pain score | up to 12 months
  11-point Pain Numbered Rating Scale, uses 11 points from 0 to 10 to describe the intensity of pain, 0 point means no pain, points increase as pain increases, 10 points means the most severe pain. Faces pain scale-11, a score of 1-3 points shows mild pain; 4-6 points indicate m moderate pain; 7-10 points indicate severe pain. The higher the pain score, the higher the pain.
anxiety | up to 12 months
  Beck Anxiety Inventory, a total of 21 items describe anxiety symptoms and measure 21 indicators of anxiety. A score of 0-9 points means "normal", 10-18 points indicate "mild" anxiety, 19-29 indicate "moderate" anxiety, and 30-63 points indicate "severe" anxiety.
pain control satisfaction | up to 12 months
  Visual Analogue Scale, this study used Visual Analogue Scale as a scale to assess patient satisfaction with pain control. It is explained to the patient that 0 cm means no pain, 10 cm means very pain, and moving from the left to the right means the pain is higher.
sleep quality | up to 12 months
  Chinese version of Pisttsburgh Sleep Quality Index, is the Chinese version of the Pittsburgh Sleep Quality Each aspect is scored 0-3points, so the total score is 21points. The average score of 5 points is the demarcation point of sleep quality. The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Lu, Principal Investigator — National Yang-Ming Unerversity Hospital
Locations (2):
- Taiwan (2):
  - National Yang-Ming University Hospital, Yilan
  - Taiwan: Ministry of Health and Welfare, Yilan

IPD SHARING:
Plan to Share IPD: No